CLINICAL TRIAL: NCT06252675
Title: A Multicenter Phase 2 Study of Glofitamab With Pirtobrutinib for Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: Glofitamab With Pirtobrutinib for Relapsed or Refractory Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry); Adaptive Biotechnologies (Industry)
Responsible Party: Principal Investigator, Madhav Seshadri, MD, Principal Investigator, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 232516; NCI-2024-00054 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2024-01-31; First posted 2024-02-12 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — obinutuzumab; glofitamab; pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (obinutuzumab, glofitamab, pirtobrutinib) (Experimental): Participants receive obinutuzumab IV on days 1 and 2 of cycle 1 for a total of 2 doses. Participants receive glofitamab IV on days 8 and 15 of cycle 1 and day 1 of remaining cycles. Cycles repeat every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Participants receive pirtobrutinib PO once a day (QD) on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity up to Cycle 30, Day 22. Participants also undergo FDG-PET/CT at screening, after every 4 cycles through cycle 13 and then after every 6 cycles. Participants will undergo a bone marrow biopsy and aspiration at cycle 13 and blood sample collection throughout study and a tissue biopsy at relapse or progression.
  Interventions: Biological: Obinutuzumab; Biological: Glofitamab; Drug: Pirtobrutinib; Procedure: Tumor Imaging; Procedure: Biospecimen Collection; Device: ClonoSeq Assay; Procedure: Bone Marrow Biopsy

INTERVENTIONS:
Biological: Obinutuzumab — Given intravenously (IV)
  Other Names: Anti-CD20 Monoclonal Antibody R715; huMAB(CD20); RO5072759
Biological: Glofitamab — Given IV
  Other Names: Anti-CD3 Bispecific Monoclonal Antibody RO7082859; RO7082859
Drug: Pirtobrutinib — Given Orally (PO)
  Other Names: LOXO-305
Procedure: Tumor Imaging — Undergo regular care imaging/scans
  Other Names: FDG-PET; Computed Tomography (CT)
Procedure: Biospecimen Collection — Blood and tissue samples
  Other Names: Biological Sample Collection
Device: ClonoSeq Assay — ClonoSEQ is an FDA-cleared, Clinical Laboratory Improvement Amendments of 1988 (CLIA)-validated measure used to determine minimal residual disease (MRD). This helps uncover how much, if any, cancer remains in your body during and after treatment.
  Other Names: ClonoSeq
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration.
  Other Names: Biopsy of Bone Marrow

SUMMARY:
This phase II trial tests the safety and effectiveness of glofitamab given in combination with pirtobrutinib in treating patients with mantle cell lymphoma that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Glofitamab and obinutuzumab are monoclonal antibodies that may interfere with the ability of cancer cells to grow and spread. Obinutuzumab may also reduce the risk of immune-related conditions from treatment. Pirtobrutinib is in a class of medications called kinase inhibitors. It works by blocking the action of the protein that signals cancer cells to multiply. Giving glofitamab in combination with pirtobrutinib may be safe, tolerable and/or effective in treating patients with relapsed or refractory mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the safety and tolerability of the combination of glofitamab and pirtobrutinib in the first six participants enrolled.

II. To evaluate the preliminary efficacy of glofitamab and pirtobrutinib in participants with relapsed or refractory mantle cell lymphoma (MCL) as measured by complete response rate.

SECONDARY OBJECTIVES:

I. To evaluate the preliminary efficacy of glofitamab and pirtobrutinib in participants with relapsed or refractory MCL as measured by progression-free survival and overall survival.

II. To characterize the magnitude and duration of anti-tumor activity by objective response rate and duration of response.

III. To characterize the safety and tolerability of the combination of glofitamab and pirtobrutinib.

IV. To evaluate the preliminary efficacy of glofitamab and pirtobrutinib in participants with relapsed or refractory MCL as measured by complete response without measurable disease (CRMRD-) rate.

V. To evaluate the time-to-complete response without measurable residual disease (CRMRD-).

VI. To evaluate the treatment-free interval among participants who discontinue treatment following CRMRD- status.

EXPLORATORY OBJECTIVES:

I. To explore associations between baseline tumor characteristics including genetic (e.g. mutations in BTK) and immune profiles (e.g. expression of co-inhibitory receptors and T cell phenotypes) and outcomes in participants administered the combination of glofitamab and pirtobrutinib.

II. To explore the effects of the combination of glofitamab and pirtobrutinib on pharmacodynamic markers relating to drug mechanism (e.g. emergence of clones with mutations conferring resistance to the study combination).

III. To estimate the quality of life of participants during therapy with glofitamab and pirtobrutinib.

IV. To explore time-to-CRMRD- during therapy with glofitamab and pirtobrutinib.

OUTLINE:

Participants receive study treatments until the absence of disease progression or unacceptable toxicity. Participants may also have a bone marrow biopsy and aspiration at cycle 13 and plasma and blood samples collected throughout study for correlative research. Additionally, participants may undergo a tissue biopsy at relapse or progression. Participants are followed for 30 days after treatment discontinuation for safety. Participants who discontinue treatment due to complete response (CR) with undetectable MRD will complete in-person visits through the end of study visit, 94 weeks from start of treatment. Participants who discontinue treatment for any reason other than CR will be followed every 3 months for up to 94 weeks from start of treatment, until death, loss to follow up, study termination, or participant withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of signing the informed consent form.
* Have a life expectancy (in the opinion of the investigator) of at least 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky > 60%).
* History of previously treated MCL meeting the following criteria: Relapsed after or failed to respond to at least one prior line of systemic therapy including anti-CD20 monoclonal antibody and alkylator-containing chemotherapy.
* At least one bi-dimensionally measurable nodal lesion ( > 1.5 cm in its largest dimension by PET/CT scan), or at least one bi-dimensionally measurable extranodal lesion ( > 1.0 cm in its largest dimension by PET/CT scan) and FDG-avid.
* Availability of leftover tissue from the time of progression for pathology confirmation and correlative studies. Note: Formalin fixed paraffin embedded blocks are preferred. If blocks are not available, 12-15 slides containing unstained, serial sections are acceptable.
* Hemoglobin ≥ 9 g/dL (Independent of transfusions and within 7 days prior to screening assessment).
* Absolute neutrophil count >= 1.0 x 10^9/L (Independent of growth factor support and within 7 days prior to screening assessment).
* Platelets ≥ 75 x 10^9/L or >= 50 x 10^9/L if due to bone marrow involvement (Independent of transfusions and within 7 days prior to screening assessment, and independent of growth factor support and within 7 days prior to screening assessment). If the patient is cytopenic there should be no evidence of myelodysplasia orhypoplastic bone marrow.
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (or ≤ 3 x ULN for participants with Gilbert syndrome, or <= 3 x ULN if due to underlying lymphoma).
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase (SGOT)) <= 2.5 X institutional upper limit of normal.
* Alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase (SGPT)) <= 2.5 X institutional upper limit of normal.
* Creatinine clearance >= 50 mL/min (by Cockcroft-Gault formula).
* Activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) <= 1.5 x ULN.
* Prothrombin (PT) or (international normalized ratio (INR) <= 1.5 x ULN.
* In women of childbearing potential, negative serum pregnancy test within 7 days prior to study treatment and either abstinence or use of highly effective contraception methods from the time of screening for at least 18 months after pre-treatment with obinutuzumab, 2 months after the final dose of glofitamab, 1 month after last dose of pirtobrutinib, 3 months after the final dose of tocilizumab (if applicable), whichever is longer. Women of childbearing potential should not donate oocytes for 1 month after last dose of pirtobrutinib.
* For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm, with female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 3 months after pre-treatment with obinutuzumab, 2 months after the final dose of glofitamab, 28 days after last dose of pirtobrutinib, 3 months after the final dose of tocilizumab (if applicable), whichever is longer.
* Willing and capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
* Participants with prior treatment-related adverse events (AEs) must have recovered to grade <= 1 with the exception of alopecia and grade 2 peripheral neuropathy.
* Participants must be able to swallow oral medications.
* Participants with positive hepatitis B core antibody (anti-HBc) and negative hepatitis B surface antigen (HBsAg) require a negative hepatitis B polymerase chain reaction (PCR) evaluation before initiating study treatment on cycle 1 day 1. Participants with positive anti-HBc antibody are required to receive prophylactic antiviral therapy with lamivudine, tenofovir, or entecavir for the duration of treatment and for at least 6 months following the end of study treatment. Hepatitis B PCR should be repeated as clinically indicated.
* Individuals with a history of hepatitis C virus (HCV) infection must have been treated and cured. For individuals with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

Exclusion Criteria:

* Pregnant, or intention of becoming pregnant during the study or within 18 months after treatment with obinutuzumab or 2 months after the last dose of glofitamab, or 3 months after treatment with tocilizumab, whichever is longer; and 1 month after the last dose of pirtobrutinib.
* Participants should avoid chest-feeding until at least 1 week after discontinuing pirtobrutinib.
* Have received the following treatments/procedures prior to study entry:

  * Participants who experienced a major bleeding event or grade ≥ 3 arrhythmia on prior treatment with a BTK inhibitor. NOTE: Major bleeding is defined as bleeding having one or more of the following features: potentially life-threatening bleeding with signs or symptoms of hemodynamic compromise; bleeding associated with a decrease in the hemoglobin level of at least 2g per deciliter; or bleeding in a critical area or organ (e.g., retroperitoneal, intraarticular, pericardial, epidural, or intracranial bleeding or intramuscular bleeding with compartment syndrome)
  * Participants who discontinued a covalent BTK inhibitor due to disease progression or relapse. NOTE: Participants who discontinued covalent BTK inhibitor therapy due to intolerance will not be excluded. Covalent BTK inhibitor intolerance is defined as:

    * Any grade 3 or higher non-hematologic toxicity, except a major bleeding event or grade >= 3 arrhythmia which are exclusion criteria
    * Any grade 1 or higher non-hematologic toxicity that lasted longer than 7 days or recurred
    * Any grade 4 hematologic toxicity
    * Neutropenic fever
    * Discontinuation due to drug interaction/expected toxicity with resolution of prior covalent BTK inhibitor-related toxicities
  * Any CD20/CD3-directed bispecific antibodies for treatment of lymphoma
  * Allogeneic stem cell transplant (SCT) within 6 months or on active immunosuppression or active graft versus host disease (GVHD)
  * Solid organ transplantation
* Have received the following treatments/procedures prior to study entry whether investigational or approved, within the respective time periods prior to initiation of study treatment:

  * Radiotherapy within 2 weeks prior to the first dose of study treatment. Note: If participants have received radiotherapy within 4 weeks prior to the first study treatment administration, participants must have at least one measurable lesion outside of the radiation field
  * Autologous SCT within 90 days prior to first study treatment
  * Chimeric antigen receptor (CAR) T-cell therapy within 60 days before first study treatment or if ongoing toxicity ≥ grade 2
  * Use of monoclonal antibodies or antibody-drug conjugates within 4 weeks prior to first study treatment
  * Use of radioimmunoconjugates within 12 weeks prior to first study treatment
  * Systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks or five half-lives (whichever is shorter) prior to first dose of study treatment. Note: Systemic corticosteroid treatment . 10 mg/day prednisone or equivalent and inhaled corticosteroids are permitted. Administration of acute, low-dose, systemic immunosuppressant medications (e.g., single dose of dexamethasone for nausea or B symptoms) is permitted. The use of mineralocorticoids for management of orthostatic hypotension and corticosteroids for management of adrenal insufficiency is permitted
  * Live, attenuated vaccine within 4 weeks before first dose of study treatment, or in whom it is anticipated that such a live attenuated vaccine will be required during the study period or within 5 months after the final dose of study treatment
* Evidence of active central nervous system (CNS) lymphoma or leptomeningeal infiltration
* Current or history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease. Note: Participants with a history of stroke who have not experienced a stroke or transient ischemic attack within the past 2 years and have no residual neurologic deficits, as judged by the investigator, are allowed
* Active second malignancy unless the patient is in remission and has a life expectancy > 2 years.
* Major surgical procedure (under general anesthesia) within 30 days of day 1 of protocol therapy. Note: If a patient had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibody therapy (or recombinant antibody-related fusion proteins).
* History of autoimmune disease, including but not limited to myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain- Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis Note: Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone, participants with a history of disease-related immune thrombocytopenic purpura or autoimmune hemolytic anemia, and participants with a history of type I diabetes mellitus who are well controlled (defined as a screening glycosylated hemoglobin (hemoglobin A1c) ≤ 8% and no urinary ketoacidosis) may be eligible for this study. Investigators should consult the sponsor-investigator.
* Significant or extensive history of cardiovascular disease such as New York Heart Association class III or IV or objective class C or D cardiac disease, myocardial infarction within the previous 6 months, unstable arrhythmia, or unstable angina or acute coronary syndrome within the past 2 months prior to start of study treatment (cycle 1 day 1 (C1D1)), uncontrolled or symptomatic arrhythmias, and/or documented left ventricular ejection fraction (LVEF) by any method of ≤ 40% in the 12 months prior to start of study treatment (C1D1)
* Prolongation of the QTc for heart rate using Fridericia's Formula (QTcF) > 470 msec. Note: Correction of QTc for underlying bundle branch block is permissible.
* Significant pulmonary disease that is expected to interfere with therapy.
* History of confirmed progressive multifocal leukoencephalopathy (PML).
* Known active infection (including Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)), or reactivation of a latent infection, whether bacterial, viral (including, but not limited to, Epstein-Barr virus (EBV), cytomegalovirus (CMV), hepatitis B and hepatitis C), fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 4 weeks (relating to the completion of the course of antibiotics) prior to first study treatment administration.
* Participants requiring therapeutic anticoagulation with warfarin or another vitamin K antagonist.
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH).
* Participants who have tested positive for human immunodeficiency virus (HIV) are excluded due to risk of opportunistic infections with both HIV and BTK inhibitors. For participants with unknown HIV status, HIV testing will be performed at screening and result must be negative for enrollment.
* Participants with a history of bleeding diathesis.
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of the study drug.
* A known hypersensitivity to any of the excipients of pirtobrutinib or to any of the intended study medications.
* Participants requiring ongoing therapy with strong Cytochrome P450, family 3, subfamily A (CYP3A) inhibitors or inducers will be excluded. For participants who are able to discontinue therapy with a strong CYP3A modulator, a washout period of at least 5 half-lives is required before beginning study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with high grade, treatment-emergent adverse events (AEs) | Approximately 2 weeks
  The severity of the toxicities will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. AEs and clinically significant laboratory abnormalities meeting grade 3 4 or 5 will be summarized by maximum intensity and relationship to study drug for the first 6 participants from the initiation of the study drug combination (Cycle 2 Day 8 (C2D8)) through the end of cycle 2 (Cycle 2 Day 21 (C2D21)), approximately 14 days.
Proportion of participants with Complete Response (CR) | Up to 94 weeks
  CR will be defined as the proportion of treated participants who experience a CR per Lugano criteria among evaluable participants. The Lugano classification recommends the Deauville five-point scale for reporting response by Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET)/Computerized tomography (CT): (1) no uptake or no residual uptake (when used interim) (2) slight uptake, but below blood pool (mediastinum) (3) uptake above mediastinal, but below or equal to uptake in the liver (4) uptake slightly to moderately higher than liver (5) markedly increased uptake or any new lesion (on response evaluation) from cycle 5 Day 1 through the follow-up period up to 94 weeks.
Proportion of participants with reported Cytokine-release syndrome (CRS) | Approximately 2 weeks
  The proportion of participants with a diagnosed incident of CRS for the first 6 participants from the initiation of the study drug combination (Cycle 2 Day 8 (C2D8)) through the end of cycle 2 (Cycle 2 Day 21 (C2D21)), approximately 14 days, and graded according to the American Society of Transplantation and Cellular Therapy (ASTCT) criteria will be reported.
Proportion of participants with immune effector cell-associated neurotoxicity syndrome (ICANS) | Approximately 2 weeks
  The proportion of participants with a diagnosed incident of ICANS for the first 6 participants from the initiation of the study drug combination (Cycle 2 Day 8 (C2D8)) through the end of cycle 2 (Cycle 2 Day 21 (C2D21)), approximately 14 days, and graded according to the American Society of Transplantation and Cellular Therapy (ASTCT) criteria will be reported.
Proportion of participants with reported Hemophagocytic lymphohistiocytosis (HLH) | Approximately 2 weeks
  The proportion of participants with a diagnosed incident of HLH for the first 6 participants from the initiation of the study drug combination (Cycle 2 Day 8 (C2D8)) through the end of cycle 2 (Cycle 2 Day 21 (C2D21)), approximately 14 days, and graded according to the American Society of Transplantation and Cellular Therapy (ASTCT) criteria will be reported.

SECONDARY OUTCOMES:
Median Progression-free survival (PFS) | Up to 94 weeks
  PFS will be defined as the time that elapses between initiation of trial therapy and the earlier of the day of first documented disease progression or death from any cause. Progression is defined by Lugano criteria of (1) new or increased adenopathy; an individual node must be abnormal with: (a) longest transverse diameter (LDi) >1.5 cm AND (2) splenic volume increase (3) new or larger non-measured lesions (4) recurrent previously resolved lesions (5) new extranodal lesion >1 cm in any axis (new lesions <1 cm in any axis are included if these are "unequivocally attributable" to lymphoma) (6) a new node >1.5 cm in any axis . PFS will be summarized using Kaplan-Meier method.
Median Overall Survival (OS) | Up to 94 weeks
  OS will be defined as the time that elapses between the initiation of trial therapy and the date of death from any cause for all evaluable participants. OS will be summarized using Kaplan-Meier method.
Objective Response Rate (ORR) | Up to 94 weeks
  OR will be defined as the proportion of treated participants who experience an objective response (CR or partial response (PR) per Lugano criteria) among evaluable participants.
Duration of response (DOR) | Up to 94 weeks
  DOR will be defined as the time that elapses between the day of first documented response to trial therapy (CR or PR, whichever is first recorded) and subsequent disease progression.
Proportion of participants with complete response without measurable disease (CRMRD) | At cycle 13, day 1 (a cycle is 21 days)
  CRMRD will be defined as the achievement of =< 1 x 10-6 malignant cells in peripheral blood, as assessed by ClonoSEQ assay in a participant who meets all other criteria for CR.
Median Time to CRMRD | Up to 94 weeks
  Time to CRMRD will calculate the time that elapses between the initiation of trial therapy and the day of first documented CRMRD and summarized using Kaplan-Meier method.
Median Treatment-free interval | Up to 94 weeks
  Treatment-free interval will be defined as the time that elapses from CRMRD status to the time of recurrence and summarized using Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Seshadri, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, Davis, Davis, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No